CLINICAL TRIAL: NCT06222645
Title: Comparison Between Fluorescenceimaging With Photoplethysmography （PPG） and Indocyaningreen (ICG) for Tissue Perfusion in Gastrointestinal Resections
Brief Title: PPG vs. ICG in Gastrointestinal Resections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Collaborators: Shandong Linglong Yingcheng Hospital (Network); High-Tech Clinic Beloostrov (Unknown)
Responsible Party: Principal Investigator, Xuan Qiu, Principal Investigator, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: spbuippg001
Record Dates: First submitted 2023-12-21; First posted 2024-01-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Anastomosis; Perfusion; Postoperative Complications; Gastrointestinal Neoplasms; Gastric Cancer (GC); Colorectal Cancer
Keywords: Photoplethysmography; Indocyanine Green; Fluorescence Imaging; Anastomotic Leak; Gastrointestinal Surgery; Tissue Perfusion; Intraoperative Monitoring
MeSH Terms: conditions — Postoperative Complications; Gastrointestinal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: This study employs a randomized, parallel-group design. Participants are randomly allocated to one of two distinct intraoperative assessment arms:
  1. iPPG Arm: Perfusion assessment is guided solely by the investigational Imaging Photoplethysmography (iPPG) system.
  2. ICG Arm: Perfusion assessment is guided by the standard Indocyanine Green (ICG) fluorescence imaging. The evaluation within this arm is comprehensive, encompassing both qualitative assessment (real-time visual interpretation of the angiogram by the surgeon) and quantitative analysis (software-based kinetics of the fluorescence intensity).
  The primary comparative analysis will benchmark the outcomes from the iPPG arm against those from the combined qualitative and quantitative assessments in the ICG arm.
Masking Description: For the purpose of objective quantitative analysis, all recorded imaging sequences (iPPG and ICG) will be anonymized and randomized. A dedicated data analyst, who is masked to the group identity (iPPG vs. ICG) and clinical outcomes of each sequence, will then process this dataset to extract the perfusion parameters (e.g., iPPG waveform amplitude, ICG time-to-peak). The surgical team remains unblinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indocyanine green (ICG) imaging system (Active Comparator): Participants in this arm undergo intraoperative tissue perfusion assessment guided by the standard Indocyanine Green (ICG) fluorescence imaging. This involves intravenous ICG injection. Perfusion is evaluated comprehensively through both qualitative (surgeon's visual interpretation) and quantitative (computer-based analysis of fluorescence kinetics, e.g., time-to-peak) methods. This arm represents the current standard of care.
  Interventions: Drug: ICG fluorescence imaging technology; Device: Imaging Photoplethysmography System
- imaging photoplethysmography (iPPG) (Experimental): Participants in this arm undergo intraoperative tissue perfusion assessment guided by the investigational Imaging Photoplethysmography (iPPG) system. This non-contact, camera-based technique detects microvascular blood volume changes without requiring exogenous contrast agents. The surgical team uses the real-time iPPG perfusion maps to evaluate anastomotic viability and guide surgical decisions.
  Interventions: Drug: ICG fluorescence imaging technology; Device: Imaging Photoplethysmography System

INTERVENTIONS:
Drug: ICG fluorescence imaging technology — This intervention involves the intravenous injection of the fluorescent contrast agent Indocyanine Green (ICG), followed by imaging with a near-infrared fluorescence camera system. Upon illumination with near-infrared light, ICG in the bloodstream fluoresces, allowing for real-time visualization of blood flow and tissue perfusion (qualitative assessment). Additionally, the fluorescence intensity over time can be recorded for subsequent quantitative analysis of perfusion kinetics.
  Other Names: ICG Imaging; ICG Angiography; Near-Infrared Fluorescence Imaging
Device: Imaging Photoplethysmography System — Imaging photoplethysmography is a non-contact, camera-based optical imaging technique. This investigational system operates by detecting subtle modulations in optical signals associated with pulsatile blood volume changes in microvascular tissue. It utilizes a conventional video camera to capture these signals and generates real-time tissue perfusion maps without the need for any exogenous contrast agents. The system is designed to provide intraoperative guidance for assessing tissue viability during gastrointestinal anastomoses.
  Other Names: iPPG; PPG Imaging

SUMMARY:
This randomized controlled trial compares a novel optical technique against the standard of care for assessing tissue perfusion in gastrointestinal surgery. Participants are randomized to receive either intraoperative imaging photoplethysmography (iPPG) or indocyanine green (ICG) fluorescence imaging. In the ICG group, the fluorescence data are comprehensively analyzed in two distinct ways: (1) Qualitative Assessment: real-time visual interpretation of the angiogram flow by the operating surgeon; and (2) Quantitative Assessment: software-based analysis of fluorescence kinetics (e.g., time-to-peak, maximum intensity) to generate objective perfusion parameters. The study aims to determine the agreement between the iPPG-based evaluations and both the qualitative and quantitative dimensions of the ICG standard.

DETAILED DESCRIPTION:
This randomized, parallel-group clinical study aims to compare two intraoperative imaging strategies for assessing tissue perfusion in a spectrum of gastrointestinal anastomoses, including both gastro-intestinal and entero-enteric reconstructions. The primary objective is to evaluate the diagnostic performance and clinical utility of a novel, non-contact optical technique-imaging photoplethysmography (iPPG)-against the current clinical standard, indocyanine green (ICG) fluorescence imaging.

Eligible and consented patients will be randomly assigned to one of two arms. The iPPG Arm will undergo perfusion evaluation solely using the investigational iPPG system. This method leverages a conventional video camera to detect pulsatile blood volume changes in microvascular tissue, offering a non-invasive, contrast-agent-free approach to perfusion assessment. The ICG Arm will be assessed using the standard fluorescence imaging protocol. A key feature of the study design is the pre-specified, comprehensive analysis within the ICG arm, which will incorporate both a qualitative assessment (the surgeon's real-time visual interpretation of the angiogram) and a quantitative analysis (computer-based calculation of fluorescence kinetics parameters, such as time-to-peak and inflow slope).

The study is designed to provide a head-to-head comparison of the two guiding strategies. Outcomes from the iPPG-guided arm will be systematically benchmarked against those from the ICG-guided arm. Furthermore, the internal comparison between qualitative and quantitative assessments within the ICG arm will yield valuable insights into the optimal methodology for interpreting perfusion data in clinical practice. This design allows for the evaluation of iPPG not only as a potential alternative to ICG but also for the refinement of the standard itself.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years).
* Scheduled to undergo an elective gastrointestinal resection requiring a primary gastro-intestinal or entero-enteric anastomosis.
* Able to understand and provide written informed consent.

Exclusion Criteria:

* Known hypersensitivity or allergy to indocyanine green (ICG), iodine, or any component of the ICG formulation.
* Severe hepatic impairment (e.g., Child-Pugh Class C).
* Pregnancy or lactation.
* Emergency surgery.
* Inability to comply with the study protocol or follow-up schedule in the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Anastomotic Leak | 30 days postoperatively
  Comparison of the rate of clinically significant anastomotic leak between the iPPG-guided group and the ICG-guided group. Anastomotic leak is defined as a full-thickness defect requiring radiological, endoscopic, or surgical intervention, as confirmed by an independent clinical events committee within 30 days postoperatively.
Incidence of Anastomotic Leak: Qualitative vs Quantitative ICG Assessment | 30 days postoperatively
  Comparison of the rate of clinically significant anastomotic leak between patients whose intraoperative assessment was based on qualitative ICG imaging (surgeon's visual interpretation) versus those assessed with quantitative ICG parameters (software-based kinetic analysis). Anastomotic leak is defined as a full-thickness gastrointestinal defect requiring postoperative radiological, endoscopic, or surgical intervention, as confirmed by an independent adjudication committee. This analysis will be performed specifically within the cohort of patients randomized to the ICG arm.

SECONDARY OUTCOMES:
Diagnostic Performance for Predicting Anastomotic Leak | he perfusion assessment is performed intraoperatively. The outcome (anastomotic leak) is assessed at 30 days postoperatively.
  To evaluate and compare the diagnostic accuracy of the intraoperative iPPG assessment versus the standard ICG assessment (including both qualitative and quantitative methods) in predicting the occurrence of a postoperative anastomotic leak. The perfusion assessment during surgery will be dichotomized as 'inadequate' or 'adequate'. Diagnostic performance metrics including Sensitivity, Specificity, Positive Predictive Value (PPV), Negative Predictive Value (NPV), and the Area Under the Receiver Operating Characteristic Curve (AUC-ROC) will be calculated for each modality against the clinical outcome of anastomotic leak.
Rate of Anastomotic Revision Based on Perfusion Assessment | Intraoperative (Measured immediately following the perfusion assessment of the initially constructed anastomosis)
  To quantify and compare the immediate impact of perfusion assessment on surgical decision-making by recording the frequency at which the operating surgeon decides to revise the anastomosis (i.e., resect and re-anastomose the bowel segment) based solely on the intraoperative findings of either iPPG or ICG imaging. The revision rate will be calculated as the proportion of patients in each arm (iPPG and ICG) for whom the anastomosis was revised due to perceived inadequate perfusion.
Overall Postoperative Complication Rate | 30 days postoperatively
  To comprehensively evaluate and compare the overall postoperative morbidity between the iPPG-guided group and the ICG-guided group. All complications occurring within 30 days after surgery will be recorded and graded according to the Clavien-Dindo classification system. This standardized system categorizes complications based on the level of intervention required for management, ranging from Grade I (any deviation from the normal postoperative course not requiring pharmacological/surgical intervention) to Grade V (death). The comparison will focus on the incidence of complications of Grade II and above.
Rate of Re-intervention | 30 days postoperatively
  To compare the incidence of unplanned, procedure-related re-interventions between the iPPG-guided and ICG-guided groups. A re-intervention is defined as any subsequent surgical, endoscopic, or radiology-guided invasive procedure required to manage a complication related to the initial gastrointestinal resection and anastomosis (e.g., control of bleeding, drainage of an intra-abdominal collection, or repair of an anastomotic leak). Planned, staged procedures are excluded. The rate is calculated as the proportion of patients in each group undergoing at least one such re-intervention.

OTHER OUTCOMES:
Surgeon Confidence Score | Intraoperative (Assessed immediately after perfusion evaluation and before fascial closure)
  To quantify the surgeon's confidence in the adequacy of the anastomotic perfusion following the intraoperative assessment. Immediately after evaluating the perfusion with the assigned modality (iPPG or ICG) and before abdominal closure, the primary surgeon will rate their confidence on an 11-point numerical rating scale, ranging from 0 (no confidence in anastomotic viability) to 10 (absolute confidence in anastomotic viability). The mean confidence scores will be compared between the two study arms.
Time from Imaging to Decision | Intraoperative (Measured for each anastomosis assessment event)
  To compare the workflow efficiency between the iPPG and ICG assessment modalities. This measure records the time elapsed from the moment a clear, interpretable perfusion image is first available on the display to the moment the surgeon verbally communicates the final decision regarding the anastomosis (e.g., "proceed as is," "revise anastomosis," "create stoma"). The time is recorded in seconds for each assessed anastomosis.

CONTACTS AND LOCATIONS:
Locations (3):
- Shandong Linglong Yingcheng Hospital, Yantai, Shandong, China
- Russia (2):
  - High-Tech Clinic Beloostrov, Saint Petersburg, Leningradskaya Oblast'
  - Department of Faculty Surgery, Saint Petersburg State University, Saint Petersburg, Leningradskaya Oblast'

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR